CLINICAL TRIAL: NCT04295018
Title: A Phase # Study Evaluating Safety and Efficacy of C-CAR088 Treatment in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA-directed CAR-T Cells Treatment in Subjects With r/r Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0203-007
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR088 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-BCMA gene
  Interventions: Drug: C-CAR088

INTERVENTIONS:
Drug: C-CAR088 — Autologous BCMA-directed CAR-T cells, single infusion intravenously at a target dose of 1.0-9.0 x 10^6 anti-BCMA CAR+T cells/kg. Other Name: CBM.BCMA Chimeric Antigen Receptor T cell.

SUMMARY:
This is a single-center, non-randomized study to evaluate the safety and efficacy of C-CAR088 in relapsed or refractory multiple myeloma patients.

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Apheresis, Baseline, Pre-Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), C-CAR088 infusion and Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female;
2. The patient volunteered to participate in the study, and he or his legal guardian signed the Informed Consent;
3. Patients with a clear diagnosis of relapsed or refractory multiple myeloma
4. The patient have one or more measurable multiple myeloma lesion, must include one of the following conditions:

   * Serum M protein≥1.0 g/dL(10g/L)
   * Urine M protein≥200 mg/24h
   * Serum free light chain(sFLC): κ/λ FLC ratio is abnormal and affected FLC ≥10mg / dL
5. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination;
6. At least 2 weeks from monoclonal antibody therapy prior to CAR T cell therapy.
7. ECOG scores 0 - 1;
8. Good cardiac and pulmonary organ function;
9. Expected survival time > 12 weeks;.
10. Female subjects of childbearing age must have a negative urine / blood pregnancy test within 7 days before cell therapy and not be in lactation; female or male subjects of childbearing age need to take effective contraception throughout the study.

Exclusion Criteria:

1. Have a history of allergy to cellular products;
2. Laboratory testing occurs when: including but not limited to, serum total bilirubin ≥1.5mg / dl; serum ALT or AST is 2.5 times higher than the upper limit of normal value; serum creatinine ≥2.0mg / dl; hemoglobin <80g / L; absolute neutrophil count <1000 / mm3 or dependent on GCSF or Other growth factors can maintain the centriole count ≥1000 / mm²; platelet count <50000 / mm³ or the above level can be maintained due to platelet transfusion;
3. Presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or any heart function Grade 3 (moderate) or Grade 4 (severe) heart disease (according to the New York Heart Association Function Classification method: NYHA); patients with a history of myocardial infarction, cardiac angioplasty or stent implantation, unstable angina pectoris or other clinically significant heart disease within 12 months before enrollment;
4. A history of craniocerebral trauma, consciousness disorder, epilepsy, severe cerebral ischemia or hemorrhagic disease;
5. Need to use any anticoagulant (except aspirin);
6. Patients requiring urgent treatment due to tumor progression or spinal cord compression;
7. Patients with CNS metastasis or symptoms of CNS involvement;
8. After allogeneic hematopoietic stem cell transplantation;
9. Plasma cell leukemia;
10. Patients with autoimmune diseases, immunodeficiency, or other immunosuppressive agents;
11. Uncontrolled active infection;
12. Have used any CAR T cell products or other genetically modified T cell therapy before;
13. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV infected persons;
14. Have a history of alcoholism, drug addiction and mental illness;
15. Participated in any other clinical trial within 1 months;
16. The investigators believe that there are other circumstances that are not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The Incidence of adverse events (TEAEs) within 30 days after intravenous infusion of C-CAR088 | 30 days

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
  ORR(including sCR / CR / VGPR / PR, based on IMWG 2016 efficacy evaluation criteria)
Progression free survival (PFS) | 6 months#12 months
  PFS(based on IMWG 2016 efficacy evaluation criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qu X, An G, Sui W, Wang T, Zhang X, Yang J, Zhang Y, Zhang L, Zhu D, Huang J, Zhu S, Yao X, Li J, Zheng C, Zhu K, Wei Y, Lv X, Lan L, Yao Y, Zhou D, Lu P, Qiu L, Li J. Phase 1 study of C-CAR088, a novel humanized anti-BCMA CAR T-cell therapy in relapsed/refractory multiple myeloma. J Immunother Cancer. 2022 Sep;10(9):e005145. doi: 10.1136/jitc-2022-005145. PMID 36100310